CLINICAL TRIAL: NCT04705480
Title: Pregabalin vs. Gabapentin on Reducing Opioid Usage in Trauma Patients
Brief Title: Pregabalin vs. Gabapentin on Reducing Opioid Usage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CAMC Health System (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Principal Investigator, Nancy Payne, Investigator, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-718
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Analgesics; Gabapentin; Injuries; Narcotics; Pain; Trauma
Keywords: Pregabalin , ,; Gabapentin; Opioid Pain Medication Use; Trauma; Opioid Usage Reduction
MeSH Terms: conditions — Wounds and Injuries; Pain | interventions — Pregabalin; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pregabalin (Experimental): Patients will receive 50 mg every 8 hours without dose titration. Patients with CrCl < 60mL/min will receive same dose given q12 hours. The q12 hour regimen may be increased to q8 hours if CrCl increases above 60mL/min during the 7 days study period or until discharge (if < 7 days post-enrollment).
  Interventions: Drug: Pregabalin 50mg
- Gabapentin (Experimental): Patients will receive 300 mg PO every 8 hours without dose titration. Patients with CrCl < 60mL/min will receive same dose given q12 hours. The q12 hour regimen may be increased to q8 hours if CrCl increases above 60mL/min during the 7 days study period or until discharge (if < 7 days post-enrollment).
  Interventions: Drug: Gabapentin 300mg
- Neither Pregabalin nor Gabapentin (Active Comparator): Patients will receive neither Pregabalin nor Gabapentin
  Interventions: Drug: Neither Pregabalin nor Gabapentin

INTERVENTIONS:
Drug: Pregabalin 50mg — Patients will receive 50 mg every 8 hours without dose titration. Patients with CrCl < 60mL/min will receive same dose given q12 hours. The q12 hour regimen may be increased to q8 hours if CrCl increases above 60mL/min during the 7 days study period or until discharge (if < 7 days post-enrollment).
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Gabapentin 300mg — Patients will receive 300 mg PO every 8 hours without dose titration. Patients with CrCl < 60mL/min will receive same dose given q12 hours. The q12 hour regimen may be increased to q8 hours if CrCl increases above 60mL/min during the 7 days study period or until discharge (if < 7 days post-enrollment).
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Neither Pregabalin nor Gabapentin — Patients will receive neither Pregabalin nor Gabapentin.
  Arms: Neither Pregabalin nor Gabapentin

SUMMARY:
This is a single-center, randomized, open-label, Phase 4 clinical trial investigating the efficacy of multiple-dose administrations of Pregabalin or Gabapentin in combination with traditional opioid pain medications to decrease the amount of opioid pain medication usage in single-system orthopedic trauma patients.

DETAILED DESCRIPTION:
Patients included in this trial were admitted under the care of the Trauma Nurse Practitioners (TNPs) who lead management of these patients. The TNP service is a 24/7 model where TNPs admit and manage patients under the trauma attending doctors from patient arrival in the emergency department until discharge, unless a higher level of care is indicated. The TNP patient census was monitored to identify new admissions who met the study criteria. Eligibility for participation was determined based on pre-established inclusion and exclusion criteria . Over the course of the trial, three changes were made to the eligibility criteria. To increase enrollment, the inclusion age range was revised from 18-70 years to 18 years and older. Additionally, the enrollment window was adjusted from 24 hours to 36 hours to facilitate the inclusion of patients admitted over the weekend. Receipt of a peripheral nerve block was also added to the exclusion criteria due to its potential to influence reported pain levels.

Patients included in the study were divided into 3 groups: pregabalin, gabapentin, and a control group receiving neither treatment. An SPSS algorithm using simple randomization was employed to generate a randomization list and assign patients to one of three groups. A sample size of 70 patients per study group (total of 210 patients) including 10% attrition was targeted. The sample size was determined based on Cohen's d formula using a power of 80%, a medium effect size indicating a 69% difference between groups. Effect sizes were calculated for planned comparisons (pregabalin vs. gabapentin, pregabalin vs. neither pregabalin nor gabapentin, gabapentin vs. neither pregabalin nor gabapentin) using t-statistics. An interim analysis was conducted after enrollment reached approximately 25% of the projected sample size to evaluate the study progress.

Enrollment and consenting of participants were performed by the research coordinators. Upon obtaining informed consent, participants were randomized sequentially to one of the three study arms by the coordinators, using the pre-generated randomization list. Enrolled patients were informed of their study arm and the TNP's initiated study drugs accordingly. Participants were followed throughout their hospital stay and remained in the study for a duration of seven days or until discharge, whichever occurred first. Patients underwent no additional cost for participating in the study as both pregabalin and gabapentin were frequently used as adjunct analgesia in this patient population at the study institution. Standard of care remained the same regardless of study participation. Patients were removed from the study if they were transferred to a higher level of care requiring a different service line.

For dosing purposes, patients with creatinine clearance (CrCl) greater than 60 ml/min received 50 mg of pregabalin every 8 hours in the pregabalin group or 300 mg of gabapentin every 8 hours in the gabapentin group. Those with CrCl less than or equal to 60ml/min received the same dose given every 12 hours, and the regimen was changed to every 8 hours if their CrCl increased above 60ml/min while enrolled. Creatine clearance was monitored daily during hospital course with dosage adjustments as necessary.

For this study, pain scores documented by nursing staff when patients requested additional pain medications were included. Pain scores were based upon a standard Numeric Rating Scale (0 = "no pain", 10 = "worst pain imaginable"). Patients who were already using prescription narcotics were eligible to participate and were continued on their home regimens as deemed necessary by providers. Adjunct non-opioid analgesia was administered at the discretion of the managing service. In-hospital narcotic exposure was ascertained by examining total amount of narotics administered in oral Morphine Milligram Equivalents (MME).

Data were collected via patient chart review and from the institution's trauma registry. Baseline patient characteristics extracted included age, gender, body mass index (BMI), days of enrollment, time from enrollment to first study drug administration, presence of rib fracture, timestamp of surgical intervention if applicable, prescription narcotics upon admission and comorbidities. Primary outcome measures included daily opioid intake during enrollment. Secondary outcomes included daily non-opioid analgesic intake, documented pain scores, post-enrollment complications (unplanned ICU admission or intubation), and daily incentive spirometry values for those with rib fractures. Additionally, adverse events such as somnolence, dizziness, fatigue, ataxia, tremor, amnesia, etc. were also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Nurse Practitioner service admissions
2. 18 years of age or older
3. Patients enrolled within 36 hours of admission
4. Anticipated duration of hospitalization > 24 hours from time of consent
5. Active order(s) for opioids in place at the time of enrollment

Exclusion Criteria:

1. Clinician discretion based on patient care management
2. Intubated patients
3. Patients with epidural
4. Patients with pregabalin/gabapentin as home medications
5. Patients receiving pregabalin/gabapentin upon admission
6. Traumatic brain injury patients
7. CrCl<30ml/min or on HD
8. Unable to take enteral medications
9. On Patient Controlled Analgesia (PCA)
10. Patients with complicated wound closure
11. History of epilepsy
12. Documented history of substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charleston Area Medical Center"s Level 1 Trauma Center, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fabbri A, Voza A, Riccardi A, Serra S, Iaco F; Study and Research Center of the Italian Society of Emergency Medicine (SIMEU). The Pain Management of Trauma Patients in the Emergency Department. J Clin Med. 2023 May 5;12(9):3289. doi: 10.3390/jcm12093289. PMID 37176729
- [Background] Ling W, Mooney L, Hillhouse M. Prescription opioid abuse, pain and addiction: clinical issues and implications. Drug Alcohol Rev. 2011 May;30(3):300-5. doi: 10.1111/j.1465-3362.2010.00271.x. PMID 21545561
- [Background] Florence C, Luo F, Rice K. The economic burden of opioid use disorder and fatal opioid overdose in the United States, 2017. Drug Alcohol Depend. 2021 Jan 1;218:108350. doi: 10.1016/j.drugalcdep.2020.108350. Epub 2020 Oct 27. PMID 33121867
- [Background] Ramirez MF, Kamdar BB, Cata JP. Optimizing Perioperative Use of Opioids: A Multimodal Approach. Curr Anesthesiol Rep. 2020 Dec;10(4):404-415. doi: 10.1007/s40140-020-00413-6. Epub 2020 Sep 7. PMID 33281504
- [Background] Simpson JC, Bao X, Agarwala A. Pain Management in Enhanced Recovery after Surgery (ERAS) Protocols. Clin Colon Rectal Surg. 2019 Mar;32(2):121-128. doi: 10.1055/s-0038-1676477. Epub 2019 Feb 28. PMID 30833861
- [Background] Ahmadi A, Bazargan-Hejazi S, Heidari Zadie Z, Euasobhon P, Ketumarn P, Karbasfrushan A, Amini-Saman J, Mohammadi R. Pain management in trauma: A review study. J Inj Violence Res. 2016 Jul;8(2):89-98. doi: 10.5249/jivr.v8i2.707. Epub 2016 Jul 7. PMID 27414816
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Background] Chin KK, Carroll I, Desai K, Asch S, Seto T, McDonald KM, Curtin C, Hernandez-Boussard T. Integrating Adjuvant Analgesics into Perioperative Pain Practice: Results from an Academic Medical Center. Pain Med. 2020 Jan 1;21(1):161-170. doi: 10.1093/pm/pnz053. PMID 30933284
- [Background] Arumugam S, Lau CS, Chamberlain RS. Use of preoperative gabapentin significantly reduces postoperative opioid consumption: a meta-analysis. J Pain Res. 2016 Sep 12;9:631-40. doi: 10.2147/JPR.S112626. eCollection 2016. PMID 27672340
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Hah J, Mackey SC, Schmidt P, McCue R, Humphreys K, Trafton J, Efron B, Clay D, Sharifzadeh Y, Ruchelli G, Goodman S, Huddleston J, Maloney WJ, Dirbas FM, Shrager J, Costouros JG, Curtin C, Carroll I. Effect of Perioperative Gabapentin on Postoperative Pain Resolution and Opioid Cessation in a Mixed Surgical Cohort: A Randomized Clinical Trial. JAMA Surg. 2018 Apr 1;153(4):303-311. doi: 10.1001/jamasurg.2017.4915. PMID 29238824
- [Background] Campbell R, Khuong JN, Liu Z, Borg C, Jackson S, Ramson DM, Kok J, Douglas N, Penny-Dimri JC, Perry LA. Perioperative gabapentinoid use lowers short-term opioid consumption following lower limb arthroplasty: Systematic review and meta-analysis. J Opioid Manag. 2021 May-Jun;17(3):251-272. doi: 10.5055/jom.2021.0635. PMID 34259336
- [Background] Markman J, Resnick M, Greenberg S, Katz N, Yang R, Scavone J, Whalen E, Gregorian G, Parsons B, Knapp L. Efficacy of pregabalin in post-traumatic peripheral neuropathic pain: a randomized, double-blind, placebo-controlled phase 3 trial. J Neurol. 2018 Dec;265(12):2815-2824. doi: 10.1007/s00415-018-9063-9. Epub 2018 Sep 21. PMID 30242745
- [Background] Gordh TE, Stubhaug A, Jensen TS, Arner S, Biber B, Boivie J, Mannheimer C, Kalliomaki J, Kalso E. Gabapentin in traumatic nerve injury pain: a randomized, double-blind, placebo-controlled, cross-over, multi-center study. Pain. 2008 Aug 31;138(2):255-266. doi: 10.1016/j.pain.2007.12.011. Epub 2008 Feb 6. PMID 18258368
- [Background] Moore RA, Straube S, Wiffen PJ, Derry S, McQuay HJ. Pregabalin for acute and chronic pain in adults. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007076. doi: 10.1002/14651858.CD007076.pub2. PMID 19588419
- [Background] Bockbrader HN, Wesche D, Miller R, Chapel S, Janiczek N, Burger P. A comparison of the pharmacokinetics and pharmacodynamics of pregabalin and gabapentin. Clin Pharmacokinet. 2010 Oct;49(10):661-9. doi: 10.2165/11536200-000000000-00000. PMID 20818832
- [Background] Evoy KE, Sadrameli S, Contreras J, Covvey JR, Peckham AM, Morrison MD. Abuse and Misuse of Pregabalin and Gabapentin: A Systematic Review Update. Drugs. 2021 Jan;81(1):125-156. doi: 10.1007/s40265-020-01432-7. PMID 33215352
- [Background] Dalsgaard H, Kim Peder Dalhoff, Heerfordt IM. A review of the addictive potential of pregabalin and gabapentin. Adverse Drug React Bull. 2024;347(1):1347-1350. doi:https://doi.org/10.1097/fad.0000000000000076
- [Background] Kuehn BM. Growing Role of Gabapentin in Opioid-Related Overdoses Highlights Misuse Potential and Off-label Prescribing Practices. JAMA. 2022 Oct 4;328(13):1283-1285. doi: 10.1001/jama.2022.13659. PMID 36069924
- [Background] Hahn J, Jo Y, Yoo SH, Shin J, Yu YM, Ah YM. Risk of major adverse events associated with gabapentinoid and opioid combination therapy: A systematic review and meta-analysis. Front Pharmacol. 2022 Oct 11;13:1009950. doi: 10.3389/fphar.2022.1009950. eCollection 2022. PMID 36304170
- [Background] Kharasch ED, Clark JD, Kheterpal S. Perioperative Gabapentinoids: Deflating the Bubble. Anesthesiology. 2020 Aug;133(2):251-254. doi: 10.1097/ALN.0000000000003394. No abstract available. PMID 32667153
- [Background] Patel AS, Abrecht CR, Urman RD. Gabapentinoid Use in Perioperative Care and Current Controversies. Curr Pain Headache Rep. 2022 Feb;26(2):139-144. doi: 10.1007/s11916-022-01012-2. Epub 2022 Jan 27. PMID 35084656
- [Background] Verret M, Lauzier F, Zarychanski R, Perron C, Savard X, Pinard AM, Leblanc G, Cossi MJ, Neveu X, Turgeon AF; Canadian Perioperative Anesthesia Clinical Trials (PACT) Group. Perioperative Use of Gabapentinoids for the Management of Postoperative Acute Pain: A Systematic Review and Meta-analysis. Anesthesiology. 2020 Aug;133(2):265-279. doi: 10.1097/ALN.0000000000003428. PMID 32667154
- See also: Center for Disease Control and Prevention. Drug overdose mortality by state. Center for Disease Control and Prevention. Published 2022. — http://www.cdc.gov
- See also: Centers for Disease Control and Prevention. About Prescription Opioids. Overdose Prevention. Published May 8, 2024 — http://www.cdc.gov/overdose-prevention/about/prescription-opioids.html
- See also: American College of Surgeons. ACS Trauma Quality Programs Best Practices Guidelines for Acute Pain Management in Trauma Patients.; 2020 — http://www.facs.org/media/exob3dwk/acute_pain_guidelines.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a tertiary, academic Level I trauma center located in the southeastern region of the United States between 2021-2024. Patients included in this trial were admitted under the care of the Trauma Nurse Practitioners (TNPs) who lead management of these patients. Screening for eligibility based on inclusion and exclusion criteria , enrollment and consenting of participants were performed by the research coordinators.
Period: Overall Study
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
Started | 43 | 33 | 33
Completed | 38 | 33 | 30
Not Completed | 5 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Decision to discharge before intervention | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin | Total
Number analyzed (Participants) | 38 | 33 | 30 | 101
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [48 to 73] | 63 [51 to 71] | 72 [57 to 74] | 61 [48 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 23 | 70
  Male | 12 | 12 | 7 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38 | 33 | 30 | 101
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m²] | 30 [28 to 34] | 30 [27 to 38] | 28 [25 to 31] | 30 [27 to 34]
Days of enrollment [Median (Inter-Quartile Range); unit: days] | 2 [1 to 5] | 3 [1 to 6] | 4 [2 to 6] | 3 [1 to 6]
Patients with rib fracture [Count of Participants; unit: Participants] | 3 | 2 | 3 | 8
Time from enrollment to first dose of study drug [Median (Inter-Quartile Range); unit: hours] | 4 [2 to 7] | 2 [1 to 4] | 0 [0 to 0] | 3 [1 to 6]
Patients underwent surgery [Count of Participants; unit: Participants] | 34 | 28 | 26 | 88
Opioids as home medication [Count of Participants; unit: Participants] | 2 | 0 | 3 | 5
Pre-existing Cardiovascular Disease [Count of Participants; unit: Participants] | 25 | 21 | 25 | 71
Pre-existing Diabetes [Count of Participants; unit: Participants] | 5 | 9 | 9 | 23
Pre-existing Smoker [Count of Participants; unit: Participants] | 9 | 6 | 5 | 20
Pre-existing Psychiatric [Count of Participants; unit: Participants] | 5 | 8 | 0 | 13
Pre-existing Pulmonary [Count of Participants; unit: Participants] | 1 | 1 | 4 | 6
Pre-existing Hematologic [Count of Participants; unit: Participants] | 2 | 0 | 3 | 5
Pre-existing Autoimmune [Count of Participants; unit: Participants] | 1 | 0 | 2 | 3
Pre-existing Neurological [Count of Participants; unit: Participants] | 1 | 2 | 0 | 3
Pre-existing Gastrointestinal [Count of Participants; unit: Participants] | 0 | 2 | 0 | 2
Pre-existing Malignancy [Count of Participants; unit: Participants] | 0 | 1 | 0 | 1
Pre-existing Other [Count of Participants; unit: Participants] | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Opioid Usage
Description: To determine if adding multiple doses of pregabalin or gabapentin upon admission will reduce opioid usage administered in oral Morphine Milligram Equivalents in trauma patients.
Time Frame: First 7 days post-enrollment or until discharge, if discharge < 7 days post-enrollment
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
Number analyzed (Participants) | 38 | 33 | 30
MME | 69.5 [35 to 115] | 81 [30 to 150] | 66.3 [45 to 120.8]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Other — The study sought to assess if adding multiple doses of pregabalin or gabapentin upon admission will reduce opioid usage in trauma patients. No specific assessment of inferiority or superiority was done; p = 0.687, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pregabalin vs Neither Pregabalin Nor Gabapentin; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.557, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gabapentin vs Neither Pregabalin Nor Gabapentin; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.601, ANCOVA; Rank transformation was applied to account this for nonparametric outcome while adjusting for significantly different psychiatric comorbidities

2. Secondary Outcome: Difference in Initial and Last Incentive Spirometry Values
Description: To compare the difference between the initial and last documented incentive spirometry values (mL) among patients in each of the study groups who have at least 1 rib fracture.
Time Frame: Initial and last incentive spirometry, with an approximate duration of 7days or discharge; if discharge < 7 days post-enrollment.
Population: The number in each arm does not match the number in the arms of the overall study as this outcomes measure pertains to those with rib fracture only.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
Number analyzed (Participants) | 3 | 2 | 3
mL | 400 [300 to 500] | 0 [0 to 0] | 250 [250 to 250]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Other; p = 0.346, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pregabalin vs Neither Pregabalin Nor Gabapentin; Test type: Other; p = 0.233, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gabapentin vs Neither Pregabalin Nor Gabapentin; Test type: Other; p = 0.145, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Rate of Intubation
Description: To compare the proportion of patients requiring intubation among the study groups.
Time Frame: First 7 days post-enrollment or until discharge, if discharge < 7 days post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
Number analyzed (Participants) | 38 | 33 | 30
Participants | 0 | 2 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Chi-squared
Statistical Analysis 2: Comparison: Pregabalin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Chi-squared
Statistical Analysis 3: Comparison: Gabapentin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Regression, Logistic; This was applied to adjust for significantly different psychiatric comorbidities

4. Secondary Outcome: Pain Control
Description: To assess effectiveness of pain control in each arm based on the average Numeric Pain Rating Scale score per 24 hours. This scale is a 10 point numeric scale that ranges from 0 that represents "no pain" to 10 which indicates the "worst pain imaginable."
Time Frame: First 7 days post-enrolment or until discharge, if discharge < 7 days post-enrollment
Measure: Median (Inter-Quartile Range); unit: Average score on numeric pain scale/day
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
Number analyzed (Participants) | 38 | 33 | 30
Average score on numeric pain scale/day | 6.4 [6.0 to 7.0] | 6.2 [5.8 to 7.0] | 6.2 [5.8 to 6.6]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pregabalin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gabapentin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, ANCOVA; [statistical method as in outcome 1, analysis 3]

5. Secondary Outcome: Hospital Length of Stay
Description: To evaluate the differences among the study arms with respect to hospital length of stay (days).
Time Frame: First 7 days post-enrollment or until discharge, if discharge < 7 days post-enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
Number analyzed (Participants) | 38 | 33 | 30
days | 3.0 [2.0 to 5.6] | 4.0 [2.0 to 6.8] | 4.3 [3.0 to 7.0]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pregabalin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Gabapentin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, ANCOVA; [statistical method as in outcome 1, analysis 3]

6. Secondary Outcome: Rate of Unplanned ICU Admission
Description: To evaluate the differences among the study arms with respect to proportion of unplanned ICU admission.
Time Frame: First 7 days post-enrollment or until discharge, if discharge < 7 days post-enrollment
Population: While enrolled, no patients in the pregabalin or neither group required ICU admission or intubation, however, these events occurred in 2 patients (6.1%) in the gabapentin group. These unplanned ICU upgrades were not due to the study medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
Number analyzed (Participants) | 38 | 33 | 30
Participants | 0 | 2 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Chi-squared
Statistical Analysis 2: Comparison: Pregabalin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Chi-squared
Statistical Analysis 3: Comparison: Gabapentin vs Neither Pregabalin Nor Gabapentin; Test type: Other — No specific assessment of inferiority or superiority was done; p < 0.05, Regression, Logistic; This was applied to adjust for significantly different psychiatric comorbidities

ADVERSE EVENTS:
Time Frame: Up to 7 days or discharge, whichever occurred first
Description: Study coordinators monitored charts for any adverse events post enrollment for 7 days or until discharge, whichever occurred first. These were reported to the PI and classified as serious or not, and reported to the IRB accordingly. Most were felt to be unrelated to study drugs. Only those reported as dizziness, somnolence or confusion were felt to possibly be related and study medications were stopped. All adverse events resolved prior to discharge.
Arm/Group | Pregabalin | Gabapentin | Neither Pregabalin Nor Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/38 | 3/33 | 3/30
Other Adverse Events (participants affected / at risk) | 1/38 | 2/33 | 4/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=38) | Gabapentin (N=33) | Neither Pregabalin Nor Gabapentin (N=30)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
hallucination or confusion (General disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
post surgical complication (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pneumatosis of colon requiring surgery (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=38) | Gabapentin (N=33) | Neither Pregabalin Nor Gabapentin (N=30)
buccal ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
dizziness and/or somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The estimated sample size was not attained due to organizational implementations of specified multi-modal regimens. The limited sample size may have rendered the study underpowered to detect significant effects and constrained the generalizability of the study findings. Inconsistences existed in gabapentinoids being initiated perioperative versus post-operatively. Pain scores were only collected at time of opioid medication requests not comprehensively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT04705480/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT04705480/ICF_001.pdf